CLINICAL TRIAL: NCT05639530
Title: A Dose Escalation Phase I Clinical Study to Evaluate the Tolerability and Safety of IBI333 in Subjects With Neovascular Age-related Macular Degeneration (nAMD)
Brief Title: A Dose Escalation Study of IBI333 in Subjects With Neovascular Age-related Macular Degeneration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CIBI333A101
Record Dates: First submitted 2022-11-14; First posted 2022-12-06 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Neovascular Age-related Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- :treated with different doses of single intravitreal injections of IBI333 (Experimental): Biological: IBI333 Dose 1 IBI333 of single IVT injections，
  Biological: IBI333 Dose 2 IBI333 of single IVT injections
  Interventions: Biological: IBI333
- treated with different doses of multiple intravitreal injections of IBI333 (Experimental): Biological: IBI333 Dose 3 IBI333 of multiple IVT injections，
  Biological: IBI333 Dose 4 IBI333 of multiple IVT injections
  Interventions: Biological: IBI333

INTERVENTIONS:
Biological: IBI333 — Intravitreal injection of IBI333

SUMMARY:
This study is designed for multi-center, open-label, dose escalation phase I trial to evaluate the safety and tolerability of a single and multiple intravitreal injection of IBI333 in subjects with neovascular age-related macular degeneration (nAMD).

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to sign informed consent form and comply with visit and study procedures per protocol.
2. Male or female patients ≥ 50 yrs. of age.
3. Active CNV lesions secondary to neovascular AMD.
4. BCVA score of 19-78 letters using ETDRS charts in the study eye.
5. Female subjects of childbearing age or male subjects with childbearing age female partner agree to take effective contraceptive measures from the screening period to 6 months after the end of treatment.

Exclusion Criteria:

1. Concomitant diseases that may cause subjects fail to respond to the treatment or confuse the interpretation of the study results;
2. Tractional retinal detachment, pre-retinal fibrosis, vitreomacular traction, or epiretinal membrane involving the fovea or disrupting the macular structure in the study eye;
3. Active ocular or periocular inflammation/infection in either eye;
4. Prior any treatment of following in the study eye:

   1. Anti-VEGF therapy within 90 days prior to screening;
   2. Intraocular glucocorticoid injection within 180 days prior to screening;
   3. Laser photocoagulation or photodynamic therapy within 90 days prior to screening;
   4. Intraocular surgery within 90 days prior to screening;
   5. Laser posterior capsulotomy, laser trabeculectomy or laser peripheral iridectomy within 30 days prior to screening;
5. Glycated hemoglobin (HbA1c) > 8% within 28 days prior to screening;
6. Uncontrolled hypertension (defined as systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg);
7. Systemic administration of steroids within 30 days prior to screening;
8. Systemic administration of anti-VEGF drugs within 90 days prior to screening;
9. History of severe hypersensitivity/allergic to active ingredients or any excipients of the study drug, or fluorescein and povidone iodine;
10. Participated in any clinical study of any other drug within 90 days prior to enrollment, or attempted to participate in other drug trials during the study;
11. Other conditions unsuitable for enrollment judged by investigators.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2023-12-07 (Actual); Study Completion 2024-04-23 (Actual)

PRIMARY OUTCOMES:
Safety and tolerance indicators | Through study completion, a maximum of 24 weeks
  1. Incidence, relatedness and severity of all adverse events (AE), treatment emergent adverse events (TEAE) and serious adverse events (SAE);
  2. Incidence of dose limiting toxicity;

SECONDARY OUTCOMES:
The area under the curve (AUC) of serum concentration of the drug after the administration. | Through study completion, a maximum of 24 weeks
Maximum concentration (Cmax) of the drug after the administration. | Through study completion, a maximum of 24 weeks
Time at which maximum concentration (Tmax) occurs for the drug after the administration. | Through study completion, a maximum of 24 weeks
The half-life (t1/2) of drug after the administration . | Through study completion, a maximum of 24 weeks
Number of participants with anti-drug antibodies or neutralizing antibodies . | Through study completion, a maximum of 24 weeks
Changes of BCVA measured by ETDRS chart from baseline. | Through study completion, a maximum of 24 weeks
Changes of CST measured by spectral domain optical coherence tomography (SD-OCT) from baseline. | Through study completion, a maximum of 24 weeks
Proportion of subjects without intraretinal or subretinal fluid on SD-OCT. | Through study completion, a maximum of 24 weeks
Change of height of pigment epithelial detachment from baseline on SD-OCT. | Through study completion, a maximum of 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No